CLINICAL TRIAL: NCT04148196
Title: Effect of Progressive Muscle Relaxation on Adaptation to Old Age and Quality of Life Among Older People in a Nursing Home: A Randomized Controlled Trial
Brief Title: The Effect of Progressive Relaxation Exercise on Adaptation to Old Age and Quality of Life.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aksaray University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Cemile KÜTMEÇ YILMAZ, Principal Investigator, Aksaray University Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019/23
Record Dates: First submitted 2019-10-30; First posted 2019-11-01 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Older People
Keywords: Older people; Adaptation; Life quality; Nursing home

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): older people's who have a Standard Mini Mental Test score of 23 and above, living in nursing homes.
- Experimental group (Experimental): Intervention group: older people's who have a Standard Mini Mental Test score of 23 and above, living in nursing homes.The researcher will perform 16 sessions of progressive relaxation exercises twice a week for 8 weeks. Each PMR exercise was conducted under the guidance of the researcher. Before and after each session of the Progressive Muscle Relaxation They will be measured heart rate and blood pressure.
  Interventions: Other: Progressive muscle relaxation exercise

INTERVENTIONS:
Other: Progressive muscle relaxation exercise — The CD on relaxation exercises developed by the Turkish Psy-chological Associationwas used.In the second of CD 27-min section; relaxation exercises are explained to the accompaniment ofrunning water sounds and verbal instructions. Progressive relaxation technique includes stretching and relaxing the bigmuscle groups (hands, arms, neck, shoulders, face, chest, abdomen,hip, feet andfingers) in the human body on purpose. When steps ofProgressive Relaxation Exercises are analyzed, it is observed thatlearning how to take correct and deep breaths is the most impor-tant step towards learning relaxation. In addition, taking correct breaths is used as a part of the exercise among all relaxation exercises.Steps of Progressive Relaxation Exercise:- breathing exercises- lower extremity exercises- upper extremity exercises- exercise of respiratory muscles. Elderly individuals will receive PMR exercise twice a week under the guidance of an investigator for eight weeks.
  Arms: Experimental group

SUMMARY:
The changes and limitations that occur in the aging process effect people's adaptation toold age. The quality of life of elderly individuals who have problems in adaptation to aging is negatively affected. This study aimed to assess the effect of effects of Progressive Muscle Relaxation on the adaptation levels and quality of life of the elderly living in nursing homes.

DETAILED DESCRIPTION:
Today, changes and developments in technology and lifestyles have lengthened average life span and increased the elderly population. The physical and cognitive changes, health problems, new roles such asbeing retired or widowed and economic losses come one after anotherfor the elderly, and this turns the old age into a period full of difficul-ties. The difficulties experienced in this period introduce problems re-lated to the adaptation of the elderly to old age. The union of the problems arising due to old age decreases the self-respect and life satisfaction of the elderly individual, and consequently, the quality of life can be negatively affected.

Adaptation is defined as the harmony built by an individual between his own needs and the expectations of the people around.It is important for people to adapt to ever-changing life events sothat they can lead happy lives.The first condition of a healthy and problem-free old age is to accept and adapt to old age.Therefore, the purposes of nursing care cover ensuring an individual's adaptation toold age and its changes, which is the last development phase of life.

Nurses can positively change people's adaptation to old age by applying simple andeconomic non-pharmacological methods that are easy to apply. The non-pharmacological methods used in this study for older people'sw included progressive muscle relaxation exercise. It is stated in the literature that progressive relaxation exercise increases the quality of life and satisfaction of elderly individuals. However, there was no study thatassessed the effect of progressive muscle relaxation exercise on adaptation to old age.

Objective: Evaluate the effects of progressive muscle relaxation on the adaptation levels older people's and quality of life of the elderly living in nursing homes.

Methodology: This is randomized clinical test. The sample was made up of 45 older people living in nursing homes (24 in control group and 21 in the experimental group). The progressive muscle relaxation technique was employed. In order to collect the data, we adopted the interview with form filling technique, using the introductory information form, Assessment Scale of Adaptation Difficulty for the Elderly (ASADE) and Nottingham Health Profile (NHP)". Blood pressure and heart rate of experimental group were measured before and after the progressive muscle relaxation intervention.

ELIGIBILITY:
Inclusion Criteria:

* 65 years and above,
* Do not have a diagnosis of dementia and psychiatric disease by the doctor and have a mini-mental test score of 23 and above,
* There is no problem with communication

Exclusion Criteria:

* Having severe hearing or perceptual deficits that impaired communication
* Having dementia, Alzheimer's disease,

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2019-11-10 (Actual); Study Completion 2019-11-25 (Actual)

PRIMARY OUTCOMES:
Standard Mini Mental Test (SMMT) | pretest of study
  SMMT evaluates cognitive status. Seniors with a SMMT score above 23 (min.0 - max. 30) were included in the study.

SECONDARY OUTCOMES:
Nottingham Health Profile | 2 months
  The health-related quality of life of elderly individuals was evaluated using the Nottingham Health Profile (NHP). he lowest and highest scores that can be obtained from each sub-dimension of the scale are 0 and 100, respectively. 0 indicates the best health status while 100 indicates the worst health status.
Assessment Scale of Adaptation Difficulty for the Elderly (ASADE) | 2 months
  The difficulties in adaptation to old age of elderly individuals were evaluated using the Assessment Scale of Adaptation Difficulty for the Elderly (ASADE). The scores obtained from the items of the scale (24 ıtems) are collected and divided by the number of questions to obtain the total score of the scale. The level of adaptation to old age decreases as the score obtained from the scale by an individual increases. ASADE total score min. 0- max. 3.

CONTACTS AND LOCATIONS:
Overall Officials: Cemile KÜTMEÇ YILMAZ, Principal Investigator — Aksaray University, Faculty of Health Science, Nursing Department, Turkey
Locations (2):
- Turkey (Türkiye) (2):
  - Cemile KÜTMEÇ YILMAZ, Merkez, Aksaray
  - Aksaray University Health Science Faculty, Aksaray

IPD SHARING:
Plan to Share IPD: No